CLINICAL TRIAL: NCT04873245
Title: Lifestyle Counseling and Medication for Adolescent Weight Management
Acronym: QUEST
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2021-29784
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Participants who qualify will be randomized to receive either intensive behavioral therapy or treatment with semaglutide plus a less intensive behavioral therapy program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intensive Behavioral Program Arm (Active Comparator): Participants randomized to this arm of the study will receive intensive behavioral therapy.
  Participants will receive 52 weekly sessions (50% in person and 50% virtual).
  Interventions: Behavioral: Intensive Behavioral Program
- Medication Arm (Active Comparator): Participants randomized to this arm of the study will receive semaglutide and will receive behavioral therapy. Behavioral therapy will consist of 12 monthly sessions (50% in person and 50% virtual).
  Interventions: Drug: Semaglutide and Behavioral Program

INTERVENTIONS:
Behavioral: Intensive Behavioral Program — Participants randomized to this group will receive intensive behavioral therapy.
  Arms: Intensive Behavioral Program Arm
Drug: Semaglutide and Behavioral Program — Participants randomized to this group will receive semaglutide and behavioral therapy.
  Arms: Medication Arm

SUMMARY:
The prevalence of adolescent severe obesity is at an all-time high in the United States and the refractory nature of this disease has led to a serious and challenging conundrum in terms of how to provide effective, safe, scalable, and durable treatments without placing undue strain on the healthcare system. Clinical practice guidelines recommend behavioral interventions as the primary strategy for all ages and classes of obesity - moderate to severe. In 2017, the U.S. Preventive Services Task Force (USPSTF) released updated screening recommendations concluding that comprehensive, intensive behavioral interventions with a total of ≥26 contact hours over a period of 2-12 months resulted in weight loss in youth with obesity, with ≥52 contact hours leading to even greater weight loss and improvements in some cardiometabolic risk factors.

However, the practicality of delivering these types of intensive behavioral services to the millions of youth with severe obesity in the U.S. is debatable not only because of the treatment-resistant nature of severe obesity, but also due to the time-commitment, acceptability, and sustainability of this approach for adolescent patients and their families along with the extensive resources required to provide these interventions. Indeed, fewer than 50% of pediatric patients referred for weight management services enroll in treatment, and high attrition rates of up to 50% have been reported in behavioral-based clinical trials and in the clinical setting. Moreover, adherence to behavioral counseling significantly diminishes over time, which too often erodes early weight loss success and ultimately derails durability. The reality of what most patients/families are able to do and the unique physiological and psychosocial features of severe obesity in adolescence do not seem to align well with the degree of intensity of behavioral interventions shown to be effective by the USPSTF. Therefore, a critical appraisal of the feasibility, effectiveness, and sustainability of the USPSTF recommendations among adolescents with severe obesity is warranted.

While behavior change is an indispensable component of any effective weight loss approach, adjunctive strategies such as pharmacotherapy may enhance outcomes in adolescents with severe obesity. Many maladaptive behaviors attributed to obesity are driven by underlying biological forces, such as increased appetite and food palatability, that are largely beyond the control of the individual. Pharmacotherapy can help facilitate behavior change by disrupting core pathophysiological processes and restoring homeostasis to the energy regulatory system, therein enabling individuals to sustain healthy behavior change. Though under-explored as a treatment for adolescent obesity, pharmacotherapy along with relatively low-intensity behavioral counseling (<26 contact hours) represents a potentially effective, durable, and safe treatment strategy. This approach may be more practical and feasible to implement on a broad scale, be preferred by patients/families, utilize fewer healthcare resources, and cost less to deliver compared to comprehensive, intensive behavioral interventions.

DETAILED DESCRIPTION:
This is a two-arm, randomized clinical trial in adolescents with severe obesity evaluating 52 weeks of intensive behavioral counseling, aligned with USPSTF recommendations (52 contact hours), vs. 52 weeks of medical management with semaglutide (glucagon-like peptide-1 receptor agonist) plus relatively low-intensity behavioral counseling (12 contact hours).

ELIGIBILITY:
Inclusion Criteria:

* Severe obesity (Body Mass Index (BMI) >/= 120% of the 95th percentile or BMI >/= 35 kg/m2)
* Age 12 to < 18 years old and Tanner stage >1

Exclusion Criteria:

* Diabetes (type 1 or 2)
* Current or recent (< 6 months prior to enrollment) use of anti-obesity medication(s) defined as orlistat, phentermine, topiramate, combination phentermine/topiramate, liraglutide (or other GLP-1RA) and/or combination naltrexone/bupropion (monotherapy use of naltrexone or bupropion is not an exclusion)
* Previous bariatric surgery
* Any history of treatment with growth hormone
* Medically-documented history of bulimia nervosa
* Major psychiatric disorder as determined by the local medical monitor
* Unstable depression requiring hospitalization within the previous 6 month
* Any history of suicide attempt
* History of suicidal ideation or self-harm within the previous 30 days
* Current pregnancy or plans to become pregnant
* ALT or AST >/= 5 times the upper limit of normal
* Creatinine > 1.2 mg/dL
* Uncontrolled hypertension as determined by the local medical monitor
* Diagnosed and medically-documented monogenic obesity
* Medically-documented history of cholelithiasis
* Untreated thyroid disorder
* Medically documented history of pancreatitis
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* Clinically significant heart disease as determined by the local medical monitor
* Personal history of malignant neoplasms within the past five years
* Hypersensitivity to any component of semaglutide

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index | 52 weeks
  The percent change in body mass index (BMI) from Baseline to Week 52 will be calculated. BMI is defined as a person's weight in kilograms divided by the square of height in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Kelly, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Delaware Clinical Research Unit, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
To be determined
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Sharing will be available 10 years after the trial has been concluded.
Access Criteria: Individuals should contact the study PI for information.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT04873245/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT04873245/ICF_001.pdf